CLINICAL TRIAL: NCT05430087
Title: The Combination of Vitamin D and Curcumin Piperine Attenuates the Disease Activity and Pro-Inflammatory Cytokines Levels in Systemic Lupus Erythematosus Patients
Brief Title: Vitamin D and Curcumin Piperine Attenuates Disease Activity and Cytokine Levels in Systemic Lupus Erythematosus Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Saiful Anwar Hospital (Other)
Responsible Party: Principal Investigator, Dr. dr. Cesarius Singgih Wahono, SpPD-KR, Rheumatologist, Rheumatology Division Department of Internal Medicine, Faculty of Medicine Universitas Brawijaya - Saiful Anwar General Hospital, Saiful Anwar Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 38/SK/UN10.F08.06/KS/2019
Record Dates: First submitted 2022-05-22; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: systemic lupus erythematosus; vitamin D; curcumin; piperine; disease activity
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Patients who fulfilled the inclusion and exclusion criteria were randomized into three parallel groups: Vitamin D + placebo (group I), Curcumin-Piperine + placebo (group II), and vitamin D + Curcumin-Piperine (group III). All patients and physicians were blinded to group assignment and treatment allocation
Who Masked: Participant, Investigator
Masking Description: All patients and physicians were blinded to group assignment and treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vitamin D + Placebo (Experimental): The first group received 400 IU cholecalciferol (Nature Plus) t.i.d (three times a day) and placebo (Saccharum lactis) t.i.d.
  Interventions: Drug: Observe the clinical outcome and inflammatory cytokines levels in patients with systemic lupus erythematosus (SLE) after being supplemented with Cholecalciferol (Vitamin D3) and Curcumin-Piperine.
- Curcumin-Piperine + Placebo (Experimental): The second group received a tablet containing curcumin (632 mg) - piperine (15,800 mg) (Bioglan) one time daily and a placebo (Saccharum lactis) t.i.d.
  Interventions: Drug: Observe the clinical outcome and inflammatory cytokines levels in patients with systemic lupus erythematosus (SLE) after being supplemented with Cholecalciferol (Vitamin D3) and Curcumin-Piperine.
- Vitamin D + Curcumin-Piperine (Experimental): The third group received 400 IU cholecalciferol (Nature Plus) t.i.d and curcumin (600 mg) - piperine (15,800 mg) (Bioglan) one time daily
  Interventions: Drug: Observe the clinical outcome and inflammatory cytokines levels in patients with systemic lupus erythematosus (SLE) after being supplemented with Cholecalciferol (Vitamin D3) and Curcumin-Piperine.

INTERVENTIONS:
Drug: Observe the clinical outcome and inflammatory cytokines levels in patients with systemic lupus erythematosus (SLE) after being supplemented with Cholecalciferol (Vitamin D3) and Curcumin-Piperine. — All patients and physicians were blinded to group assignment and treatment allocation. All subjects received the tablets for three months. All subjects were still required to consume their routine medications during the supplementation according to the disease activity. Patients were evaluated at baseline and after the end of supplementation for clinical and laboratory parameters. Adherence to therapy was assessed by monthly pill counts of returned tablets and biweekly phone calls to the patients.

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic systemic autoimmune disease with a relatively high mortality and morbidity rate, especially in developing countries such as Indonesia. In Indonesia, a previous study demonstrated that almost 71% of SLE patients experience hypovitaminosis D, with serum vitamin D 25 levels less than 30 ng/ml. Several factors contribute to the low vitamin D levels among SLE patients. Less exposure to sunlight or insufficient vitamin D intake contributes to SLE patients low vitamin D levels. Some other studies also revealed that vitamin D metabolism gene polymorphisms are also associated with patients with SLE.

Vitamin D is essential for bone health and has an essential role in immune system modulation and controlling autoimmune diseases, including SLE. Another study demonstrates that curcumin supplementation in premenopausal women and dysmenorrhea improves vitamin D levels. Despite the promising properties of curcumin in improving vitamin D biological actions, our previous study reveals that the addition of curcumin in vitamin D administration do not significantly improve the disease activity or cytokine imbalance in SLE patients. The synergistic property of curcumin with vitamin D in regulating immune cells is an open opportunity for researchers to increase the response to vitamin D3 therapy.

Several studies have reported the efficacy of vitamin D or curcumin for SLE treatment. However, none mentioned the combination of curcumin added with piperine and vitamin D3. We hypothesized that adding curcumin piperine with vitamin D3 as a complementary treatment in SLE patients would improve the clinical symptoms or cytokine balance among SLE patients. Therefore, this study aims to observe the effects of adding curcumin-piperine with vitamin D3 in clinical outcomes and cytokines levels in SLE patients with hypovitaminosis D.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic systemic autoimmune disease with a relatively high mortality and morbidity rate, especially in developing countries such as Indonesia. In Indonesia, a previous study demonstrated that almost 71% of SLE patients experience hypovitaminosis D, with serum vitamin D (25(OH)D3) levels less than 30 ng/ml. Several factors contribute to the low vitamin D levels among SLE patients. Less exposure to sunlight or insufficient vitamin D intake contributes to SLE patients' low vitamin D levels. Some other studies also revealed that vitamin D metabolism gene polymorphisms are also associated with patients with SLE.

Vitamin D is essential for bone health and has an essential role in immune system modulation and controlling autoimmune diseases, including SLE. An increase in the pro-inflammatory cytokine, such as interleukin-6 (IL-6), is found in SLE patients with hypovitaminosis D. SLE patients with hypovitaminosis D have a more severe clinical condition and disease activity. However, previous meta-analysis shows that vitamin D supplementation is effective in increasing the serum 25(OH)D levels, may improve fatigue, and is well-tolerated in patients with SLE. However, it does not seem to have significant effects in decreasing the positivity of anti-dsDNA and disease activity. Thus, another approach to enhance the effect of vitamin D to suppress the pro-inflammatory condition in SLE should be considered.

Curcumin is a phenolic compound widely found in ginger, turmeric, and curcuma plants and has the potential as an immunomodulator for the complementary treatment of SLE. Curcumin acts as an activator or inhibitor of several transcription factors that play a role in activating and differentiating Th1, Th2, Th17, and Tregs. In a previous report, curcumin synergistically interacts with vitamin D because it is also a natural ligand for the vitamin D receptor (VDR). Previous studies reveal that administering a combination of curcumin and vitamin D3 resulted in a better recovery of neuronal cells from Alzheimer's disease. Another study demonstrates that curcumin supplementation in premenopausal women and dysmenorrhea improves vitamin D levels.

Despite the promising properties of curcumin in improving vitamin D biological actions, our previous study reveals that the addition of curcumin in vitamin D administration do not significantly improve the disease activity or cytokine imbalance in SLE patients. Because of the pharmacokinetics of curcumin, this substance is poorly absorbed in the gut and has low bioavailability when administered by the oral route. Therefore, special treatment is needed to improve the bioavailability of curcumin. One of the potential strategies is adding the piperine when administering curcumin orally. Piperine can be found in plants of the Piperaceae family, including 2-7.4% of black pepper and white pepper (Piper nigrum L.). Piperine also has antioxidant, immunomodulatory, and anti-inflammatory activities. Piperine can increase the in vivo bioavailability of curcumin by inhibiting its metabolism and reducing the required dose of curcumin in the clinical setting. Piperine can also increase cell membrane permeability, thereby increasing drug absorption. Piperine binds to several areas of the enzyme to form a hydrogen bond complex with curcumin that can increase its bioavailability up to twenty times.

The synergistic property of curcumin with vitamin D in regulating immune cells is an open opportunity for researchers to increase the response to vitamin D3 therapy. Several studies have reported the efficacy of vitamin D or curcumin for SLE treatment. However, none mentioned the combination of curcumin added with piperine and vitamin D3. We hypothesized that adding curcumin piperine with vitamin D3 as a complementary treatment in SLE patients would improve the clinical symptoms or cytokine balance among SLE patients. Therefore, this study aims to observe the effects of adding curcumin-piperine with vitamin D3 in clinical outcomes and cytokines levels in SLE patients with hypovitaminosis D.

ELIGIBILITY:
Inclusion Criteria:

* SLE patients referred to the Rheumatology outpatient clinic Saiful Anwar General Hospital, Malang, Indonesia
* Had an active disease, characterized by the Mexican SLE Disease Activity Index (Mex-SLEDAI) score >3
* Had low vitamin D levels (serum vitamin D3 levels <30 ng/ml)

Exclusion Criteria:

* Pregnant or breast-feeding patients
* Took supplementations containing vitamin D or curcumin in the last three months
* Had severe liver disorders (AST or ALT levels >2.5 times of upper normal limit)
* Had impaired renal function (GFR < 25 ml/min or oliguria with urine output < 400 ml/day)
* Had other autoimmune diseases or severe infections such as tuberculosis, pneumonia, or HIV, history of renal stones, hypercalciuria, intestinal malabsorption
* Refusal to participate in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Disease Activity from the SLE patients after the Treatments | three months
  Disease activity was assessed using the Mexican SLE Disease Activity Index (Mex-SLEDAI) score, consisting of 10 simple clinical and laboratory components obtained during the examination, which the results are grouped into remission (score of 0-1), mild (score of 2-5), moderate (score of 6-9), severe (score of 10-13), and very severe (score of > 14).
Fatigue Assessment from the SLE patients after the Treatments | three months
  Fatigue assessment was done using a specific questionnaire called the Fatigue Severity Scale (FSS) score. The FSS score used in this study was a validated Indonesian version consisting of nine questions to assess fatigue, including physical functioning, vitality, emotional, social, and mental health. The items are scored on a seven point scale with 1 refers to strongly disagree and 7 refers to strongly agree. The minimum FSS score is 9 and the maximum score possible is 63, with the higher the score the greater the fatigue severity
Comparison of Cytokines Levels before and After the Treatments | three months
  We also monitor the pro-inflammatory and anti-inflammatory cytokines from the sera of SLE patients three months after the therapies
  Serum cytokine levels, including interleukin-6 (IL-6) and transforming growth factor-β (TGF-β), were measured at the baseline and three months after therapy using enzyme-linked immunosorbent assay (ELISA) by the commercially kits (Elabscience, cat number E-EL-H0102 and E-EL-0162, respectively). Both results were shown in pg/ml.

CONTACTS AND LOCATIONS:
Locations (1):
- Saiful Anwar General Hospital, Malang, East Java, Indonesia

REFERENCES:
- [Result] Hamijoyo L, Candrianita S, Rahmadi AR, Dewi S, Darmawan G, Suryajaya BS, Rainy NR, Hidayat II, Moenardi VN, Wachjudi RG. The clinical characteristics of systemic lupus erythematosus patients in Indonesia: a cohort registry from an Indonesia-based tertiary referral hospital. Lupus. 2019 Nov;28(13):1604-1609. doi: 10.1177/0961203319878499. Epub 2019 Sep 29. PMID 31566078
- [Result] Islam MA, Khandker SS, Alam SS, Kotyla P, Hassan R. Vitamin D status in patients with systemic lupus erythematosus (SLE): A systematic review and meta-analysis. Autoimmun Rev. 2019 Nov;18(11):102392. doi: 10.1016/j.autrev.2019.102392. Epub 2019 Sep 11. PMID 31520805
- [Result] Breslin LC, Magee PJ, Wallace JM, McSorley EM. An evaluation of vitamin D status in individuals with systemic lupus erythematosus. Proc Nutr Soc. 2011 Nov;70(4):399-407. doi: 10.1017/S0029665111001613. Epub 2011 Aug 24. PMID 21861947
- [Result] Ruiz-Ballesteros AI, Meza-Meza MR, Vizmanos-Lamotte B, Parra-Rojas I, de la Cruz-Mosso U. Association of Vitamin D Metabolism Gene Polymorphisms with Autoimmunity: Evidence in Population Genetic Studies. Int J Mol Sci. 2020 Dec 17;21(24):9626. doi: 10.3390/ijms21249626. PMID 33348854
- [Result] Hamza RT, Awwad KS, Ali MK, Hamed AI. Reduced serum concentrations of 25-hydroxy vitamin D in Egyptian patients with systemic lupus erythematosus: relation to disease activity. Med Sci Monit. 2011 Dec;17(12):CR711-8. doi: 10.12659/msm.882131. PMID 22129903
- [Result] Terrier B, Derian N, Schoindre Y, Chaara W, Geri G, Zahr N, Mariampillai K, Rosenzwajg M, Carpentier W, Musset L, Piette JC, Six A, Klatzmann D, Saadoun D, Patrice C, Costedoat-Chalumeau N. Restoration of regulatory and effector T cell balance and B cell homeostasis in systemic lupus erythematosus patients through vitamin D supplementation. Arthritis Res Ther. 2012 Oct 17;14(5):R221. doi: 10.1186/ar4060. PMID 23075451
- [Result] Aranow C, Kamen DL, Dall'Era M, Massarotti EM, Mackay MC, Koumpouras F, Coca A, Chatham WW, Clowse ME, Criscione-Schreiber LG, Callahan S, Goldmuntz EA, Keyes-Elstein L, Oswald M, Gregersen PK, Diamond B. Randomized, Double-Blind, Placebo-Controlled Trial of the Effect of Vitamin D3 on the Interferon Signature in Patients With Systemic Lupus Erythematosus. Arthritis Rheumatol. 2015 Jul;67(7):1848-57. doi: 10.1002/art.39108. PMID 25777546
- [Result] de Souza VA, Bastos MG, Fernandes NM, Mansur HN, Raposo NR, de Souza DM, de Andrade LC. Association of hypovitaminosis D with Systemic Lupus Erythematosus and inflammation. J Bras Nefrol. 2014 Oct-Dec;36(4):430-6. doi: 10.5935/0101-2800.20140062. English, Portuguese. PMID 25517270
- [Result] Mok CC, Birmingham DJ, Leung HW, Hebert LA, Song H, Rovin BH. Vitamin D levels in Chinese patients with systemic lupus erythematosus: relationship with disease activity, vascular risk factors and atherosclerosis. Rheumatology (Oxford). 2012 Apr;51(4):644-52. doi: 10.1093/rheumatology/ker212. Epub 2011 Jun 29. PMID 21719424
- [Result] Correa-Rodriguez M, Pocovi-Gerardino G, Callejas-Rubio JL, Rios-Fernandez R, Martin-Amada M, Cruz-Caparros MG, DelOlmo-Romero S, Ortego-Centeno N, Rueda-Medina B. Vitamin D Levels are Associated with Disease Activity and Damage Accrual in Systemic Lupus Erythematosus Patients. Biol Res Nurs. 2021 Jul;23(3):455-463. doi: 10.1177/1099800420983596. Epub 2020 Dec 30. PMID 33380211
- [Result] Zheng R, Gonzalez A, Yue J, Wu X, Qiu M, Gui L, Zhu S, Huang L. Efficacy and Safety of Vitamin D Supplementation in Patients With Systemic Lupus Erythematosus: A Meta-analysis of Randomized Controlled Trials. Am J Med Sci. 2019 Aug;358(2):104-114. doi: 10.1016/j.amjms.2019.04.020. Epub 2019 Apr 26. PMID 31331447
- [Result] Momtazi-Borojeni AA, Haftcheshmeh SM, Esmaeili SA, Johnston TP, Abdollahi E, Sahebkar A. Curcumin: A natural modulator of immune cells in systemic lupus erythematosus. Autoimmun Rev. 2018 Feb;17(2):125-135. doi: 10.1016/j.autrev.2017.11.016. Epub 2017 Nov 24. PMID 29180127
- [Result] Bartik L, Whitfield GK, Kaczmarska M, Lowmiller CL, Moffet EW, Furmick JK, Hernandez Z, Haussler CA, Haussler MR, Jurutka PW. Curcumin: a novel nutritionally derived ligand of the vitamin D receptor with implications for colon cancer chemoprevention. J Nutr Biochem. 2010 Dec;21(12):1153-61. doi: 10.1016/j.jnutbio.2009.09.012. Epub 2010 Feb 12. PMID 20153625
- [Result] Alamro AA, Alsulami EA, Almutlaq M, Alghamedi A, Alokail M, Haq SH. Therapeutic Potential of Vitamin D and Curcumin in an In Vitro Model of Alzheimer Disease. J Cent Nerv Syst Dis. 2020 May 27;12:1179573520924311. doi: 10.1177/1179573520924311. eCollection 2020. PMID 32528227
- [Result] Arabnezhad L, Mohammadifard M, Rahmani L, Majidi Z, Ferns GA, Bahrami A. Effects of curcumin supplementation on vitamin D levels in women with premenstrual syndrome and dysmenorrhea: a randomized controlled study. BMC Complement Med Ther. 2022 Jan 22;22(1):19. doi: 10.1186/s12906-022-03515-2. PMID 35065636
- [Result] Singgih Wahono C, Diah Setyorini C, Kalim H, Nurdiana N, Handono K. Effect of Curcuma xanthorrhiza Supplementation on Systemic Lupus Erythematosus Patients with Hypovitamin D Which Were Given Vitamin D3 towards Disease Activity (SLEDAI), IL-6, and TGF-beta1 Serum. Int J Rheumatol. 2017;2017:7687053. doi: 10.1155/2017/7687053. Epub 2017 Dec 28. PMID 29445400
- [Result] Liu W, Zhai Y, Heng X, Che FY, Chen W, Sun D, Zhai G. Oral bioavailability of curcumin: problems and advancements. J Drug Target. 2016 Sep;24(8):694-702. doi: 10.3109/1061186X.2016.1157883. Epub 2016 Mar 17. PMID 26942997
- [Result] Haq IU, Imran M, Nadeem M, Tufail T, Gondal TA, Mubarak MS. Piperine: A review of its biological effects. Phytother Res. 2021 Feb;35(2):680-700. doi: 10.1002/ptr.6855. Epub 2020 Sep 14. PMID 32929825
- [Result] Shoba G, Joy D, Joseph T, Majeed M, Rajendran R, Srinivas PS. Influence of piperine on the pharmacokinetics of curcumin in animals and human volunteers. Planta Med. 1998 May;64(4):353-6. doi: 10.1055/s-2006-957450. PMID 9619120
- [Result] Aringer M, Costenbader K, Daikh D, Brinks R, Mosca M, Ramsey-Goldman R, Smolen JS, Wofsy D, Boumpas DT, Kamen DL, Jayne D, Cervera R, Costedoat-Chalumeau N, Diamond B, Gladman DD, Hahn B, Hiepe F, Jacobsen S, Khanna D, Lerstrom K, Massarotti E, McCune J, Ruiz-Irastorza G, Sanchez-Guerrero J, Schneider M, Urowitz M, Bertsias G, Hoyer BF, Leuchten N, Tani C, Tedeschi SK, Touma Z, Schmajuk G, Anic B, Assan F, Chan TM, Clarke AE, Crow MK, Czirjak L, Doria A, Graninger W, Halda-Kiss B, Hasni S, Izmirly PM, Jung M, Kumanovics G, Mariette X, Padjen I, Pego-Reigosa JM, Romero-Diaz J, Rua-Figueroa Fernandez I, Seror R, Stummvoll GH, Tanaka Y, Tektonidou MG, Vasconcelos C, Vital EM, Wallace DJ, Yavuz S, Meroni PL, Fritzler MJ, Naden R, Dorner T, Johnson SR. 2019 European League Against Rheumatism/American College of Rheumatology classification criteria for systemic lupus erythematosus. Ann Rheum Dis. 2019 Sep;78(9):1151-1159. doi: 10.1136/annrheumdis-2018-214819. Epub 2019 Aug 5. PMID 31383717
- [Result] Uribe AG, Vila LM, McGwin G Jr, Sanchez ML, Reveille JD, Alarcon GS. The Systemic Lupus Activity Measure-revised, the Mexican Systemic Lupus Erythematosus Disease Activity Index (SLEDAI), and a modified SLEDAI-2K are adequate instruments to measure disease activity in systemic lupus erythematosus. J Rheumatol. 2004 Oct;31(10):1934-40. PMID 15468356
- [Result] Magro R, Saliba C, Camilleri L, Scerri C, Borg AA. Vitamin D supplementation in systemic lupus erythematosus: relationship to disease activity, fatigue and the interferon signature gene expression. BMC Rheumatol. 2021 Dec 3;5(1):53. doi: 10.1186/s41927-021-00223-1. PMID 34857051
- [Result] Karimzadeh H, Shirzadi M, Karimifar M. The effect of Vitamin D supplementation in disease activity of systemic lupus erythematosus patients with Vitamin D deficiency: A randomized clinical trial. J Res Med Sci. 2017 Jan 27;22:4. doi: 10.4103/1735-1995.199089. eCollection 2017. PMID 28400826
- [Result] Stockton KA, Kandiah DA, Paratz JD, Bennell KL. Fatigue, muscle strength and vitamin D status in women with systemic lupus erythematosus compared with healthy controls. Lupus. 2012 Mar;21(3):271-8. doi: 10.1177/0961203311425530. Epub 2011 Oct 17. PMID 22004972
- [Result] Lima GL, Paupitz J, Aikawa NE, Takayama L, Bonfa E, Pereira RM. Vitamin D Supplementation in Adolescents and Young Adults With Juvenile Systemic Lupus Erythematosus for Improvement in Disease Activity and Fatigue Scores: A Randomized, Double-Blind, Placebo-Controlled Trial. Arthritis Care Res (Hoboken). 2016 Jan;68(1):91-8. doi: 10.1002/acr.22621. PMID 25988278
- [Result] Wobke TK, Sorg BL, Steinhilber D. Vitamin D in inflammatory diseases. Front Physiol. 2014 Jul 2;5:244. doi: 10.3389/fphys.2014.00244. eCollection 2014. PMID 25071589
- [Result] Peng Y, Ao M, Dong B, Jiang Y, Yu L, Chen Z, Hu C, Xu R. Anti-Inflammatory Effects of Curcumin in the Inflammatory Diseases: Status, Limitations and Countermeasures. Drug Des Devel Ther. 2021 Nov 2;15:4503-4525. doi: 10.2147/DDDT.S327378. eCollection 2021. PMID 34754179
- [Result] Marinho A, Carvalho C, Boleixa D, Bettencourt A, Leal B, Guimaraes J, Neves E, Oliveira JC, Almeida I, Farinha F, Costa PP, Vasconcelos C, Silva BM. Vitamin D supplementation effects on FoxP3 expression in T cells and FoxP3+/IL-17A ratio and clinical course in systemic lupus erythematosus patients: a study in a Portuguese cohort. Immunol Res. 2017 Feb;65(1):197-206. doi: 10.1007/s12026-016-8829-3. PMID 27423437
- [Result] Handono K, Pratama MZ, Endharti AT, Kalim H. Treatment of low doses curcumin could modulate Th17/Treg balance specifically on CD4+ T cell cultures of systemic lupus erythematosus patients. Cent Eur J Immunol. 2015;40(4):461-9. doi: 10.5114/ceji.2015.56970. Epub 2016 Jan 15. PMID 26862311
- [Result] Guimaraes-Stabili MR, de Aquino SG, de Almeida Curylofo F, Tasso CO, Rocha FRG, de Medeiros MC, de Pizzol JP Jr, Cerri PS, Romito GA, Rossa C Jr. Systemic administration of curcumin or piperine enhances the periodontal repair: a preliminary study in rats. Clin Oral Investig. 2019 Aug;23(8):3297-3306. doi: 10.1007/s00784-018-2755-9. Epub 2018 Nov 29. PMID 30498979
- [Derived] Wahono CS, Susianti H, Hakim AL, Rosita F, Pratama MZ, Rahman PA, Anshory M. Randomised Clinical Trial Study: The Combination of Vitamin D and Curcumin Piperine Attenuates Disease Activity and Pro-inflammatory Cytokines Levels Insystemic Lupus Erythematosus Patients. Curr Rheumatol Rev. 2024;20(5):586-594. doi: 10.2174/0115733971276106231226071002. PMID 38299416